CLINICAL TRIAL: NCT03283098
Title: A Phase 1, Multiple Dose, Randomized, Double-blind, Placebo-controlled Study to Evaluate Pharmacokinetics, Safety and Tolerability of AMG 416 Administered Intravenously to Chinese Subjects With Chronic Kidney Disease on Hemodialysis
Brief Title: A Phase 1 Study to Evaluate PK, Safety and Tolerability of AMG 416
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20140197
Record Dates: First submitted 2017-08-31; First posted 2017-09-14 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Secondary hyperparathyroidism; Chronic kidney disease CKD; Intact parathyroid hormone iPTH; Hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Intervention Model Description: This is a multiple dose, double-blind, randomized, placebo-controlled clinical study conducted in Chinese subjects residing in Mainland China with chronic kidney disease receiving hemodialysis. The treatment duration will be approximately 4 weeks with a post treatment followup of 4 weeks. A dose will be given at each scheduled hemodialysis session (Dose administered three times a week for 4 weeks, for a total of 12 doses).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Intravenous (IV) administration of placebo three times a week (TIW) for 4 weeks for a total of 12 doses. Participants were followed for an additional 4 weeks.
  Interventions: Drug: Placebo
- Etelcalcetide (Experimental): 5 mg intravenous (IV) dose of etelcalcetide three times a week (TIW) for 4 weeks for a total of 12 doses. Participants were followed for an additional 4 weeks.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Etelcalcetide was supplied as a sterile, preservative-free, aqueous solution in a single-use 3 mL glass vial.
  Other Names: AMG 416
  Arms: Etelcalcetide
Drug: Placebo — Placebo supplied to match active intervention.
  Arms: Placebo

SUMMARY:
This was a multiple-dose, double-blind, randomized, placebo-controlled study. Chinese subjects residing in Mainland China with chronic kidney disease (CKD) receiving hemodialysis were randomized in a 3:1 ratio to receive 5 mg intravenous (IV) of etelcalcetide or placebo 3 times a week (TIW) for approximately 4 weeks, with a subsequent follow up period of approximately 4 weeks.

Doses were given at the end of each scheduled hemodialysis session on study days 1 through day 27 and subject participation was complete after day 55 end-of-study (EOS) procedures were performed. Doses were administered TIW for 4 weeks, for a total of 12 doses.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* Resident in Mainland China and of Chinese ancestry
* Male or female subject ≥ 18 and ≤ 70 years of age at the time of screening, with end stage renal disease receiving hemodialysis
* Subject must be receiving hemodialysis 3 times weekly for at least 3 months through a functioning permanent dialysis access prior to Day -2 and have adequate hemodialysis with a delivered Kt/V ≥ 1.2 or urea reduction ratio (URR) ≥ 65% within 4 weeks to screening. The subject's routine hemodialysis session must be of 3-4.5 hours in duration, inclusive
* Subject has stable dialysis prescription and this prescription is not anticipated to significantly change during the course of the study

Exclusion Criteria:

* Corrected calcium (calculated) level is < 2.07 mmol/L (8.3 mg/dL), and/or intact PTH level is outside the range of 31.8 - 127.3 pmol/L (300 - 1200 pg/mL)
* Female subjects who are pregnant, lactating/breastfeeding, or who plan to conceive, or breastfeed while on study through 3 months after receiving the dose of study drug
* Female subject of reproductive potential not willing to use a(n) acceptable method(s) of effective birth control during treatment with AMG 416, and for an additional 3 months after the end of treatment with AMG 416. Female subjects who have had a hysterectomy, bilateral salpingectomy, bilateral oophorectomy, bilateral tubal ligation, or who are postmenopausal are not required to use contraception. Postmenopausal is defined as:

  * Age > 55 years with cessation of menses for 12 months or more
  * Age < 55 but no spontaneous menses for at least 2 years
  * Age < 55 years and spontaneous menses within the past 1 years, but currently amenorrheic, AND with postmenopausal gonadrotropin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (<5.3 pmol/L or 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved
  * Underwent a bilateral oophorectomy
* Females of reproductive potential with a positive pregnancy test, unless medical follow-up confirms the subject is not pregnant
* Previous administration of AMG 416
* Subject has received cinacalcet within the 30 days prior to informed consent (treatment with cinacalcet is prohibited during the study)
* Subject has lost 500 mL or more of blood or plasma within 8 weeks of study drug administration or during the study period
* Anticipated or scheduled to have major surgical procedures during the study period such as kidney transplant or parathyroidectomy
* History of malignancy within 5 years before Day -2 (except non melanoma skin cancers, or cervical carcinoma in situ)
* Subject's 12-lead electrocardiogram (ECG) at screening suggests unstable arrhythmia or other cardiac abnormality that could place the subject at increased risk, based upon the Investigator's opinion
* Subject has current or history of cardiovascular conditions such as uncontrolled hypertension, symptomatic ventricular dysrhythmias, Torsades de Pointes, angina pectoris congestive heart failure (New York Heart Association Classification III or IV), myocardial infarction, coronary angioplasty, or coronary arterial bypass grafting within the past 6 months prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- China (3):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Nanjing, Jiangsu
  - Research Site, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Xing C, Chen J, Zuo L, Fang Y, Ding X, Ni Z, Kong C, Shi G, Lu H, Hellawell J, Cheng S, Sohn W. A Phase I, Multiple-Dose, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Pharmacokinetics, Safety, and Tolerability of Etelcalcetide Administered Intravenously to Chinese Patients With Chronic Kidney Disease Undergoing Hemodialysis. Clin Ther. 2021 Nov;43(11):2013-2023. doi: 10.1016/j.clinthera.2021.09.019. Epub 2021 Nov 11. PMID 34774334
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 centers in China.
Pre-assignment Details: Of the 37 subjects screened, 33 participants were randomized in a 3:1 ratio to either etelcalcetide or placebo in a double-blind manner prior to the Day 1 activities.
Groups:
- Placebo: Intravenous (IV) administration of placebo three times a week (TIW) administered at the end of dialysis for 4 weeks for a total of 12 doses (on Study Days 1, 3, 6, 8, 10, 13, 15, 17, 20, 22, 24, 27) . Participants were followed for an additional 4 weeks.
- Etelcalcetide: 5 mg intravenous (IV) dose of etelcalcetide three times a week (TIW) administered at the end of dialysis for 4 weeks for a total of 12 doses (on Study Days 1, 3, 6, 8, 10, 13, 15, 17, 20, 22, 24, 27). Participants were followed for an additional 4 weeks.
Period: Overall Study
Arm/Group | Placebo | Etelcalcetide
Started | 8 | 25
Completed | 8 | 24
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisting of all participants who received at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Etelcalcetide | Total
Number analyzed (Participants) | 8 | 25 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (12.5) | 50.2 (11.4) | 50.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 5 | 15 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 25 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 167.54 (8.17) | 164.48 (7.68) | 165.22 (7.79)
Weight [Mean (Standard Deviation); unit: kg] | 65.74 (8.45) | 67.71 (13.53) | 67.24 (12.40)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI equals a person's weight in kilograms divided by baseline height in meters squared (kg/m^2).
  kg/m^2 | 23.64 (3.03) | 24.98 (4.03) | 24.65 (3.81)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 139.25 (27.37) | 141.24 (19.39) | 140.76 (21.13)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 80.38 (13.54) | 81.68 (13.00) | 81.36 (12.93)
Intact Parathyroid Hormone (iPTH) [Mean (Standard Deviation); unit: pmol/L] | 74.10 (35.08) | 63.03 (20.10) | 65.72 (24.40)
Corrected Calcium [Mean (Standard Deviation); unit: mmol/L] | 2.57 (0.12) | 2.46 (0.20) | 2.49 (0.19)
Calcium [Mean (Standard Deviation); unit: mmol/L] | 2.57 (0.14) | 2.44 (0.22) | 2.47 (0.21)
Phosphorus [Mean (Standard Deviation); unit: mmol/L] | 2.17 (0.49) | 2.11 (0.58) | 2.13 (0.55)
Potassium [Mean (Standard Deviation); unit: mmol/L] | 4.67 (0.48) | 4.74 (0.80) | 4.72 (0.73)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: Time to Maximum Drug Concentration (Tmax) of Plasma Etelcalcetide on Days 1 and 27
Description: Tmax is the time to maximum drug concentration of plasma etelcalcetide after dosing on Days 1 and 27.
Time Frame: Days 1 and 27; PK blood sampling predialysis, and at 10, 30, 60, 90 min postdose, as well as on Day 2 and 28 between 18 and 30 hours after study drug administration
Population: Pharmacokinetic Concentration Analysis Set: all participants who received at least 1 dose of etelcalcetide and had at least 1 pharmacokinetic sample collected.
Measure: Median (Full Range); unit: hour
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 0 | 25
hour
  Day 1 |  | 0.22 [0.17 to 0.27]
  Day 27: number analyzed (Participants) | 0 | 24
  Day 27 |  | 0.22 [0.17 to 0.25]

2. Primary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of Plasma Etelcalcetide on Days 1 and 27
Description: Cmax was defined as the maximum observed plasma drug concentration measured between the time of drug administration to the beginning of the next dialysis session.
Time Frame: as for outcome 1
Population: Pharmacokinetic concentration analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 0 | 25
ng/mL
  Day 1 |  | 216 (157)
  Day 27: number analyzed (Participants) | 0 | 24
  Day 27 |  | 236 (53.7)

3. Primary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Curve From Time Zero to the Beginning of the Subsequent Hemodialysis Treatment (AUClast) of Plasma Etelcalcetide on Days 1 and 27
Description: AUClast was specifically defined in this study as the area under the concentration time curve measured from the time of drug administration to the beginning of the next dialysis session, following the first and last dose.
Time Frame: Days 1 and 27; PK blood sampling predialysis, and up to 44-50 hour postdose.at 10, 30, 60, 90 min postdose: Day 2 and 28 between 18 and 30 hours after study drug administration; Day 3 (predialysis) + Day 29
Population: Pharmacokinetic concentration analysis set
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 0 | 25
hour*ng/mL
  Day 1 |  | 1110 (311)
  Day 27: number analyzed (Participants) | 0 | 24
  Day 27 |  | 3310 (893)

4. Primary Outcome: Pharmacokinetic (PK) Parameter: Accumulation Ratio Comparing Days 1 and 27
Description: Accumulation ratio, calculated as AUClast day 27/AUClast day 1.
Time Frame: as for outcome 3
Population: Pharmacokinetic concentration analysis set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 0 | 25
ratio |  | 3.02 (0.607)

5. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: The severity of each adverse event was assessed using the NCI-CTCAE Version 4.0 according to the following:
  * Grade 1 - Mild: Asymptomatic or mild symptoms; intervention not indicated
  * Grade 2 - Moderate: Minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)
  * Grade 3 - Severe: Medically significant but not life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL
  * Grade 4 - Life-threatening
  * Grade 5 - Fatal.
  A serious AE is an AE that met one or more of the following criteria:
  * Death
  * Life-threatening
  * Required inpatient hospitalization or prolongation of an existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * A congenital anomaly/birth defect
  * Important medical events that required medical or surgical intervention to prevent one of the outcomes above.
Time Frame: Day 1 up to Day 55 (end of study)
Population: Safety Analysis set containing all participants who received at least 1 dose of investigational product (IP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 25
Participants
  All TEAEs | 7 | 25
  TEAEs Grade >= 3 | 0 | 5
  TEAEs Grade >= 4 | 0 | 1
  Serious TEAEs | 0 | 3
  TEAEs leading to study treatment discontinuation | 0 | 0
  Fatal TEAEs | 0 | 0
  Treatment-related TEAEs | 1 | 18
  Treatment-related TEAEs Grade >= 3 | 0 | 1
  Treatment-related TEAEs Grade >= 4 | 0 | 0
  Treatment-related serious TEAEs | 0 | 1
  Trt-related TEAEs leading to study trt discon | 0 | 0
  Treatment-related Fatal TEAEs | 0 | 0

6. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs) of Interest
Description: Terms were coded with Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. Narrow search criteria used for both standardized MedDRA queries (SMQ) and events of interest (EOI). One preferred term (PT) could match multiple EOIs. Infusion Reaction EOI counts included only those events which had onset day coinciding with study medication infusion and resolved on the same day or the day after onset.
Time Frame: Day 1 up to Day 55 (end of study)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 25
Participants
  Adynamic bone (EOI) | 0 | 0
  Cardiac Failure (EOI) | 0 | 0
  Convulsions (SMQ) | 0 | 0
  Fractures (EOI) | 0 | 0
  Hypersensitivity (SMQ) | 0 | 5
  Dermatitis allergic (PT) | 0 | 2
  Rash (PT) | 0 | 2
  Dermatitis (PT) | 0 | 1
  Hypocalcemia (EOI) | 0 | 11
  Blood calcium decreased (PT) | 0 | 10
  Hypocalcaemia (PT) | 0 | 2
  Hypophosphatemia (EOI) | 0 | 0
  Infusion reaction (EOI) | 0 | 1
  Hypotension (PT) | 0 | 1
  Torsade de pointes-QT prolongation (SMQ) | 0 | 0
  Ventricular tachyarrhythmias (SMQ) | 0 | 0

7. Secondary Outcome: Participants With Clinically-Significant Changes in Electrocardiograms (ECGs) From Baseline to End of Study
Description: Count of participants who exhibited a clinically significant change in the results of their 12-lead electrocardiograms (ECG) when comparing baseline to end of study ECGs.
Time Frame: Baseline is Day -2; End of Study is Day 55
Population: Safety Analysis set of participants with both a baseline and end of study ECG.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 24
Participants
  Normal Baseline / Abnormal End of Study | 0 | 2
  Abnormal Baseline / Normal End of Study | 0 | 1
  No Change in Baseline to End of Study | 8 | 21

8. Secondary Outcome: Change From Baseline to End of Study in Weight
Description: Change from baseline in weight measured at visit.
Time Frame: Day 1 up to Day 55
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 25
kg | 1.32 (0.79) | 0.76 (1.39)

9. Secondary Outcome: Change From Baseline to End of Study in Systolic and Diastolic Blood Pressures
Description: Participants remained seated for at least 10 minutes prior to measurement of predialysis heart rate and blood pressure.
Time Frame: Baseline Day 1 prior to dialysis; End of Study is Day 55
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 25
mmHg
  Systolic Blood Pressure: number analyzed (Participants) | 8 | 24
  Systolic Blood Pressure | 1.1 (15.5) | 6.1 (18.6)
  Diastolic Blood Pressure: number analyzed (Participants) | 8 | 24
  Diastolic Blood Pressure | 4.4 (9.2) | 1.5 (11.9)

10. Secondary Outcome: Baseline and Change From Baseline to End of Study in Heart Rate
Description: Participants remained seated for at least 10 minutes prior to measurement of predialysis heart rate and blood pressure.
Time Frame: Baseline Day 1 prior to dialysis; End of Study is Day 55
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 25
beats/minute
  Baseline | 79.5 (8.3) | 82.8 (13.8)
  Change from Baseline to End of Study: number analyzed (Participants) | 8 | 24
  Change from Baseline to End of Study | -2.9 (6.5) | -1.4 (8.9)

11. Secondary Outcome: Change From Baseline to End of Study in Calcium
Description: Calcium was tested at a central laboratory.
Time Frame: Baseline is Day 1 prior to dialysis; End of Study is Day 55
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 25
mmol/L | -0.10 (0.11) | -0.07 (0.12)

12. Secondary Outcome: Change From Baseline to End of Study in Corrected Calcium (cCa)
Description: Total serum calcium was corrected if the serum albumin was < 4 g/dL or 40 g/L, otherwise cCa equals total serum calcium.
  The correction formula was:
  Corrected calcium (mg/dL) = Total calcium (mg/dL) + (4 - albumin [g/dL]) * 0.8
Time Frame: Baseline is the average of Day -2 and Day 1 prior to dialysis; End of Study is Day 55
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 25
mmol/L | -0.08 (0.10) | -0.05 (0.10)

13. Secondary Outcome: Participants With Low Corrected Calcium (cCA) By Category
Description: The lowest cCA value for each participant is reported.
  Total serum calcium was corrected if the serum albumin was < 4 g/dL or 40 g/L, otherwise cCa equals total serum calcium.
  The correction formula was:
  Corrected calcium (mg/dL) = Total calcium (mg/dL) + (4 - albumin [g/dL]) * 0.8
Time Frame: Timeframes: Days 8, 15, 22, 27, 29, 34, 41, 55
Population: Safety Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 25
Participants
  Participants with cCA < 1.75 mmol/L | 0 | 0
  Participants with cCA 1.75 to < 1.87 mmol/L | 0 | 1
  Participants with cCA 1.87 to < 2.07 mmol/L | 0 | 12

14. Secondary Outcome: Baseline and Change From Baseline to End of Study in Serum Albumin
Description: Serum albumin was tested at a central laboratory.
Time Frame: Baseline is the average of Day -2 and Day 1 prior to dialysis; End of Study is Day 55
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 25
g/dL
  Baseline | 41.20 (2.37) | 39.37 (2.79)
  Change from Baseline to End of Study: number analyzed (Participants) | 8 | 24
  Change from Baseline to End of Study | -1.06 (1.81) | -0.59 (2.13)

15. Secondary Outcome: Change From Baseline to End of Study in Serum Phosphorus
Description: Serum phosphorus was tested at a central laboratory.
Time Frame: Baseline is Day 1 prior to dialysis; End of Study is Day 55
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 8 | 25
mmol/L | -0.03 (0.53) | -0.06 (0.56)

16. Secondary Outcome: Participants With Anti-etelcalcetide Antibody at Baseline and Postbaseline
Description: Participants with positive titers for antibodies to etelcalcetide could be asked to return to the clinical research unit to provide additional serum samples.
Time Frame: Baseline: Day 1 prior to dialysis. Postbaseline: Days 29 and 55 prior to dialysis
Population: Safety Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 0 | 25
Participants
  Binding antibody positive at or before baseline |  | 1
  Positive postbaseline/negative baseline |  | 0
  Transient, i.e. negative at last timepoint tested |  | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 55 (end of study)
Description: Treatment-emergent adverse events - any adverse events started on or after the first dose of investigational product (IP) up to the end of study date (Day 55).
Arm/Group | Placebo | Etelcalcetide
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/8 | 3/25
Other Adverse Events (participants affected / at risk) | 7/8 | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Etelcalcetide (N=25)
Pneumonia (Infections and infestations) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Etelcalcetide (N=25)
Arrhythmia (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 2
Eye disorder (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 0 | 10
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT03283098/SAP_000.pdf
  • Study Protocol (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT03283098/Prot_001.pdf